CLINICAL TRIAL: NCT05137093
Title: Independent Validation Study of Nighttime Scratching Quantification With Actigraphy in Adults With Atopic Dermatitis
Brief Title: Scratching Validation Study
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: SRC_NBS_GENEActiv_2019_10763
Record Dates: First submitted 2021-11-05; First posted 2021-11-30 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis
Keywords: Scratching
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy subjects
  Interventions: Device: Actigraphy Device
- Atopic dermatitis: Atopic dermatitis
  Interventions: Device: Actigraphy Device

INTERVENTIONS:
Device: Actigraphy Device — Patients will wear actigraphy device which detects scratching events.

SUMMARY:
Single center, analyst-blinded, study comparing the scratching events identified via an actigraphy scoring algorithm versus manual scoring of an overnight video recording, undertaken in a sample of 40 adult patients with atopic dermatitis and controls.

DETAILED DESCRIPTION:
The Philips scratching algorithm has been cross-validated against the gold-standard assessment of scratching. The algorithm has been used in many drug development trials, occasionally as a means of generating secondary endpoints, but most often as a means of generating exploratory endpoints. The purpose of the proposed study is therefore to validate the data generated by the scratching study compared to the gold-standard video-assessment of scratching, in an independent sample of adults with atopic dermatitis and age- and sex-matched controls

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 to 75 years, inclusive
* Be willing and able to undergo a single night of actigraphy and video monitoring overnight in a laboratory
* Be willing and able to provide informed consent
* (patients only): Diagnosed with atopic dermatitis by a clinician, following the criteria listed in Table 1.
* (patients only): IGA score ≥ 2.
* (patients only): Willing and able to use only non-medicated topical therapy (i.e., bland emollient/moisturizer) for 7 days before the overnight visit.
* Participants should be in bed a minimum of 4 hours

Exclusion Criteria:

* Any acute and/or unstable illness or medical complication which, in the opinion of a clinician, could compromise data collection and/or interpretation
* Use of any over-the-counter, prescription, or recreational drugs that may induce sleep or pruritus within 24 hours prior to overnight monitoring
* Use of any over-the-counter or prescription treatment (systemic, or topical) that could affect the course of atopic dermatitis during the study period. Key medications are listed below:

  * From 3 Months prior to overnight visit: Biological products that might have significantly affected the evaluation of atopic dermatitis condition (e.g., tumor necrosis factor inhibitors, antiimmunoglobulin IgE antibodies, anti-CD20 antibodies, anti-interleukin-4 receptor)
  * Has used systemic treatments that could affect AD within 30 days or 5 half- lives before the overnight visit. (i.e. retinoids, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and systemic corticosteroids)
  * Phototherapy treatment, laser therapy, bleach baths, tanning booths or extended sun exposure that could affect disease severity or interfere with disease assessments within 30 days before the overnight visit.
  * Use within 21 days before the overnight visit: Topical corticosteroids that were classified as super-high potency (clobetasol propionate).
  * Use within 14 days before the overnight visit: any other topical phosphodiesterase 4 (PDE4) inhibitor; Tacrolimus and pimecrolimus cream and/or ointment; Topical corticosteroids that were classified as low, medium, or high potency (e.g., fluocinonide, triamcinolone acetonide, desonide, hydrocortisone).
  * From 7 days before the overnight visit:

    * antibiotics
    * antifungal or antivirus medications
    * Antihistamines/anti-allergics: diphenhydramine, chlorpheniramine maleate, hydroxyzine)
    * Topical phosphodiesterase 4 (PDE4) inhibitor
    * Topical calcineurin inhibitors (tacrolimus and pimecrolimus cream and/or ointment)
    * Topical corticosteroids that were classified as low, medium, or high potency (e.g., fluocinonide, triamcinolone acetonide, desonide, hydrocortisone)
    * Any other topical therapy with active ingredients to treat AD or with additives that could affect AD (e.g., hyaluronic acid, urea, ceramide or filaggrin degradation products).
* Individuals clinically diagnosed with a sleep disorder who are NOT on a controlled treatment regime
* An Epworth Sleepiness Scale score of ≥11, indicating daytime hypersomnolence
* Previous diagnosis of a movement disorder, including but not limited to, restless legs syndrome, periodic limb movement disorder, Tourette's syndrome, tremor, or dystonia
* Commercial driver's license and/or high-risk occupation that could be impacted by the occurrence of daytime sleepiness
* Self-reported habitual sleep duration of <6 hours per night on average
* Shift worker, advanced/delayed circadian phase, and/or any other condition suggesting that the participant would be unable to sleep during overnight monitoring
* Self-reported pregnancy current or planned during the study
* Employee or spouse of an employee of company that designs, sells, or manufactures sleep related products and/or wearable devices (including Philips).
* (patients only): Any significant dermatological condition, other than atopic dermatitis, as determined by a clinician.
* (controls only): Any significant dermatological condition as determined by a clinician.
* Currently using medication for any skin disease/condition and could not, in the opinion of the investigator, tolerate restriction or discontinuation of the medication as required by the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy & Atopic dermatitis subjects
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and precision of the scratching algorithm with reference to the gold standard. | Through study completion, analyst review following each patient's overnight intervention/session
  Assessment of the performance of the scratching algorithm as detected by actigraphy compared to infra red video monitoring.

SECONDARY OUTCOMES:
Agreement via additional performance metrics between the scratching algorithm and the gold standard. | Through study completion, analyst review following each patient's overnight intervention/session
  Overall agreement of algorithm-determined scratching events and total duration compared to video scoring of scratching events; Other performance metrics such as Cohen's kappa and correlation between the number and duration of scratching events detected by the scratching algorithm versus video scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Clayton Sleep Institute, Maplewood, Missouri, United States

IPD SHARING:
Plan to Share IPD: No